CLINICAL TRIAL: NCT06644781
Title: A Phase 3, Multicenter, Randomized, Open-label Study of Ifinatamab Deruxtecan (I-DXd) in Subjects With Pretreated Advanced or Metastatic Esophageal Squamous Cell Carcinoma (ESCC) (IDeate-Esophageal01)
Brief Title: A Study of Ifinatamab Deruxtecan in Subjects With Pretreated Advanced or Metastatic Esophageal Squamous Cell Carcinoma (ESCC) (IDeate-Esophageal01)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS7300-202; 2023-509630-19-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; Ifinatamab deruxtecan (I-DXd); DS-7300a
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Docetaxel; Paclitaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- I-DXd (Experimental): Participants who are randomized to receive an intravenous infusion of I-DXd 12 mg/kg on Day 1 of every 21-day cycle (Q3W).
  Interventions: Drug: Ifinatamab deruxtecan
- Investigator's Choice of Chemotherapy (ICC) (Active Comparator): Participants who are randomized to receive an intravenous infusion of investigator's choice of chemotherapy (docetaxel, paclitaxel, and irinotecan HCl).
  Interventions: Drug: Docetaxel; Drug: Paclitaxel; Drug: Irinotecan hydrochloride (HCl)

INTERVENTIONS:
Drug: Ifinatamab deruxtecan — Intravenous administration
  Other Names: I-DXd
  Arms: I-DXd
Drug: Docetaxel — Intravenous administration
  Arms: Investigator's Choice of Chemotherapy (ICC)
Drug: Paclitaxel — Intravenous administration
  Arms: Investigator's Choice of Chemotherapy (ICC)
Drug: Irinotecan hydrochloride (HCl) — Intravenous administration
  Arms: Investigator's Choice of Chemotherapy (ICC)

SUMMARY:
This study is designed to assess the efficacy and safety of ifinatamab deruxtecan (I-DXd) in patients with unresectable advanced or metastatic esophageal squamous cell carcinoma (ESCC) who have experienced disease progression following treatment with a platinum-based systemic therapy and an immune checkpoint inhibitor (ICI) compared with investigator's choice of chemotherapy (ICC).

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the overall survival (OS) benefit of I-DXd compared with investigator's choice of chemotherapy (ICC).

The key secondary objectives of the study will evaluate the progression-free survival (PFS) and objective response rate (ORR) benefit of I-DXd compared with ICC.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for randomization into the study:

1. Participants aged ≥18 years (follow local regulatory requirements if the legal age of consent for study participation is >18 years old).
2. Has histologically or cytologically documented unresectable locally advanced or metastatic ESCC according to American Joint Committee on Cancer 8th edition staging system on ESCC.
3. Has disease progression post a platinum-based chemotherapy and an ICI treatment per global or local guidelines, with a maximum of 1 prior line of systemic therapy for unresectable advanced or metastatic ESCC.
4. The participant must provide adequate baseline tumor samples with sufficient quantity and quality of tumor tissue content as defined in the Laboratory Manual.
5. Has at least 1 measurable lesion on computed tomography (CT)/magnetic resonance imaging (MRI) according to RECIST v1.1 as assessed by the investigator. Measurable lesions should not be from a previously irradiated site. If the lesion at a previously irradiated site is the only selectable target lesion, a radiological assessment showing significant progression of the irradiated lesion should be provided by the investigator.
6. Has an ECOG PS of 0 or 1 within 7 days prior to Cycle 1 Day 1.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Has received prior treatment with orlotamab, enoblituzumab, or other B7-H3 targeted agents, including I-DXd.
2. Has received any topoisomerase inhibitor.
3. Has histologically or cytologically confirmed adenosquamous carcinoma subtype.
4. Is ineligible to all the chemotherapies in the comparator arm due to prior progression or intolerance.
5. Has tumor invasion into organs located adjacent to the esophageal disease site (eg, aorta or respiratory tract) at an increased risk of bleeding or fistula as assessed by the investigator.
6. Clinically active brain metastases, spinal cord compression, or leptomeningeal carcinomatosis, defined as untreated or symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive or treated brain metastases who are asymptomatic (ie, without neurologic signs or symptoms and not requiring treatment with corticosteroids or anticonvulsants) may be included in the study. Subjects must have a stable neurologic status and discontinue corticosteroid usage for at least 2 weeks prior to Screening.
7. Has any of the following within the past 6 months: cerebrovascular accident, transient ischemic attack, other arterial thromboembolic event, or pulmonary embolism.
8. Has a clinically significant corneal disease.
9. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at Screening.
10. Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses, including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the study randomization, severe asthma, chronic obstructive pulmonary disease [COPD], restrictive lung disease, pleural effusion, etc), and potential pulmonary involvement caused by any autoimmune, connective tissue, or inflammatory disorders (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis, etc), prior pneumonectomy, or requirement for supplemental oxygen.
11. Is on chronic steroid treatment (dose of 10 mg daily or more prednisone equivalent), except for low-dose inhaled steroids (for asthma/COPD), topical steroids (for mild skin conditions), or intra-articular steroid injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of randomization to the date of death due to any cause, up to approximately 54 months
  Overall Survival (OS) is defined as the time interval from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization to the date of disease progression or death due to any cause, whichever occurs first, up to approximately 54 months
  Progression-free survival (PFS) is defined as the time interval from the date of randomization to the first date of disease progression as determined by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | From the time of first dose of study drug until date of documented disease progression or death, whichever occurs first, up to approximately 54 months
  Objective response rate (ORR) is defined as the proportion of subjects with a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) as assessed by BICR per RECIST v1.1.
Duration of Response (DoR) | From the time of the first dose of study drug until the date of documented disease progression (as assessed by BICR) or death due to any cause, up to approximately 54 months
  Duration of response (DoR) is defined as the time from the date of first documentation of objective tumor response (CR or PR), which is subsequently confirmed by BICR assessment, to the first documentation of objective tumor progression (confirmed by BICR) or to death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | From the time of the first dose of study drug until the date of documented disease progression (as assessed by BICR) or death due to any cause, up to approximately 54 months
  Disease control rate (DCR) is defined as the proportion of participants with a BOR of confirmed CR, confirmed PR, or stable disease (SD) according to RECIST v1.1 and will be determined by BICR assessment review of tumor scans.
Change from baseline in European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire Score (EORTC QLQ-C30) | Baseline up to 54 months
Change from baseline in European Organisation for Research and Treatment of Cancer Esophageal Cancer Module Score (EORTC OES18) | Baseline up to 54 months
Incidence of Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, and Adverse Events of Special Interest (AESIs) | Baseline up to 54 months
  A TEAE is defined as an adverse event (AE) with a start or worsening date during the on-treatment period. A serious TEAE is defined as any untoward medical occurrence that at any dose results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event, or may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes noted. AESIs will also be assessed. AEs will be coded using MedDRA and will be graded using NCI-CTCAE v5.0.
Percentage of Participants Who Have Treatment-emergent ADA | Baseline up to 54 months
  Anti-drug antibodies (ADAs) will be measured in the plasma using a validated assay.
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) for I-DXd | Cycle 1: Before infusion (BI), end of infusion (EOI), 3 hours (hr), 6hr, 24hr, 72hr, 168hr, 336hr, 504hr postdose; Cycle 2: BI and EOI; Cycle 3: BI, EOI, and 6hr postdose; Cycle 4, 5, & every 2 cycles thereafter, up to 54 mths: BI (each cycle is 21 days)
  Plasma pharmacokinetic parameters will be assessed using noncompartmental methods.
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) for Total Anti-B7-H3 Antibody | Cycle 1: Before infusion (BI), end of infusion (EOI), 3 hours (hr), 6hr, 24hr, 72hr, 168hr, 336hr, 504hr postdose; Cycle 2: BI and EOI; Cycle 3: BI, EOI, and 6hr postdose; Cycle 4, 5, & every 2 cycles thereafter, up to 49 mths: BI (each cycle is 21 days)
  Plasma pharmacokinetic parameters will be assessed using noncompartmental methods.
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) for MAAA-1181a | Cycle 1: Before infusion (BI), end of infusion (EOI), 3 hours (hr), 6hr, 24hr, 72hr, 168hr, 336hr, 504hr postdose; Cycle 2: BI and EOI; Cycle 3: BI, EOI, and 6hr postdose; Cycle 4, 5, & every 2 cycles thereafter, up to 49 mths: BI (each cycle is 21 days)
  Plasma pharmacokinetic parameters will be assessed using noncompartmental methods.

CONTACTS AND LOCATIONS:
Locations (88):
- United States (6):
  - Providence Medical Foundation, Fullerton, California
  - Henry Ford Health System, Detroit, Michigan
  - Baptist Cancer Center, Memphis, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - John Peter Smith Hospital, Fort Worth, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
- China (20):
  - Anyang Cancer Hospital, Anyang
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Changzhou Cancer Hospital, Changzhou
  - Sichuan cancer hospital, Chengdu
  - West China Hospital Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Fujian Medical University, Hefei
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - Affiliated Hospital of Jining Medical University, Jining
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The First Affiliated Hospital of Xinxiang Medical University, Weihui
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Zhongshan Hospital Xiamen University, Xiamen
  - Subei Peoples Hospital, Yangzhou
- France (7):
  - Sainte Catherine Institut du cancer Avignon en Provence, Avignon
  - CHU Brest - Hôpital de la Cavale Blanche, Brest
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - Unité de recherche clinique ICANS, Strasbourg
  - CHU Toulouse Rangueil Service dOncologie médicale, Toulouse
- Germany (2):
  - Krankenhaus Nordwest GmbH, Frankfurt am Main
  - Hämatologisch Onkologische Praxis Eppendorf HOPE, Hamburg
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria Luigi Vanvitelli, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione Policlinico Gemelli, Rome
- Japan (17):
  - National Cancer Center Hospital, Chūōku
  - Hiroshima University Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa
  - Kagawa University Hospital, Kita-gun
  - Kobe City Hospital Organization Kobe City Medical Center General Hospital, Kobe
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Shikoku Cancer Center, Matsuyama
  - Aichi Cancer Center, Nagoya
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Saitama Cancer Center, Saitama
  - Hokkaido University Hospital, Sapporo
  - SHOWA Medical University Hospital, Shinagawa-ku
  - Keio University Hospital, Shinjuku-ku
  - The University of Osaka Hospital, Suita-shi
  - Shizuoka Cancer Center, Sunto-gun
  - Kanagawa Cancer Center, Yokohama
- Erasmus MC, Rotterdam, Netherlands
- Poland (2):
  - Zanamed Medical Clinic Sp z o o, Lublin
  - Mazowiecki Szpital Wojewódzki, Siedlce
- Romania (4):
  - Memorial Healthcare International S R L, Bucharest
  - S.C Radiotherapy Center Cluj S.R.L, Comuna Floresti
  - Centrul de Oncologie Sfantul Nectarie Craiova, Craiova
  - S.C. Sigmedical Services SRL, Suceava
- South Korea (10):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-sisouth
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (6):
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Universitario de Elche, Elche
  - Hospital Univ Regional de Málaga Hosp Civil, Málaga
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (5):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/